CLINICAL TRIAL: NCT01623193
Title: The ABC Trial - Does All-Blood Cardioplegia Prevent Blood Transfusion in Cardiac Surgery
Brief Title: The ABC Trial Does All-Blood Cardioplegia Prevent Blood Transfusion in Cardiac Surgery? A Single Centre Pilot Study
Acronym: ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pam Trenholm (Other)
Responsible Party: Sponsor-Investigator, Pam Trenholm, Principal Investigator, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABC Trial
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
Keywords: Cardioplegia; Blood transfusion; Cardiac function; Myocardial edema; Coronary artery disease; Valve disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients receive standard 4:1 cardioplegia for myocardial protection during cardiac surgery
  Interventions: Procedure: Standard cardioplegia
- Treatment (Experimental): Patients receive all-blood cardiolpegia for myocardial protection during surgery
  Interventions: Other: All-blood cardioplegia

INTERVENTIONS:
Other: All-blood cardioplegia — The treatment group will receive all-blood cardioplegia for myocardial protection during surgery
  Arms: Treatment
Procedure: Standard cardioplegia — This arm will receive standard 4:1 cardioplegia for myocardial protection during surgery
  Arms: Control

SUMMARY:
This study is a single centre pilot for a randomized trial comparing all-blood cardioplegia to more dilute 4:1 blood cardioplegia during cardiac surgery. The hypothesis is that all-blood cardioplegia will be associated with less blood transfusion and better cardiac function.

DETAILED DESCRIPTION:
This is a single centre randomized, double blind, 2 arm, parallel group pilot study comparing all-blood cardioplegia to 4:1 blood cardioplegia in patients undergoing cardiac surgery. This pilot study will support the design of a larger multicentre trial.

Subjects undergoing cardiac surgery will be randomized to receive either standard of care (4:1) or all-blood cardioplegia for myocardial protection. Neither of these cardioplegia approaches would be considered investigational. Each is in use at numerous cardiac surgical centres around the world. The cardioplegia will be delivered using the Quest medical MPS system which is a Health Canada Approved device.

Clinical endpoints will be evalauted (rate of blood transtransfusion, ICU stay, etc…). In a subset of subjects who meet specific criteria, ventricular function will be evaluated in the operating room using the CD Leycom INCA conductance catheter system.

ELIGIBILITY:
Inclusion Criteria:

* patients (male and female) undergoing isolated coronary artery bypass grafting,
* isolated aortic or mitral repair or replacement, and
* combined aortic or mitral valve repair or replacement and
* coronary bypass grafting

Exclusion Criteria:

* reoperation,
* endocarditis,
* dialysis dependant renal failure,
* pre-operative ECMO or LVAD support,
* contraindication to blood transfusion (ie. Jehovah's Witness), and
* use of irreversible anti-platelet (other than ASA) and anticoagulant agents within 48h (ie. plavix, dabigitran, GpIIb/IIIa inhibitors, argatroban).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-05-27 (Actual)

PRIMARY OUTCOMES:
Blood transfusion | 30 days
  Number of units of packed red blood cells transfused
Intra-op diastolic function | day 1
  Left ventricular chamber stiffness constant measured by conductance catheter in the operating room

SECONDARY OUTCOMES:
Mortality | 30 day
  Mortality
Duration of Ventilation | 30 day
Lentgh of stay ICU | 30 days
Length of stay - hospital | 30 day
Other blood product administration | 30 day
Hgb - arrival ICU | day 1
Hgb - prior to Discharge | 30 days
Lowest post op Hgb | 30 days
Volume of crystalloid delivered in cardioplegia | day 1
Fluid balance | 30 d
Reoperation rate for bleeding | 30 days
Inotrope score | 30 day
  Score incorporating amount and number of inotropes administered
Low output syndrome | 30 days
Troponin | 24 hours post op
Infection | 30 days
  Composite according to standardized definitions
intra-op Ventricular function | day 1
  as determined by conductance catheter

CONTACTS AND LOCATIONS:
Overall Officials: Stacy O'Blenes, MD, Principal Investigator — Dalhousie University
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada